CLINICAL TRIAL: NCT05733650
Title: Expanded Access Program (EAP) to Provide Epcoritamab (GEN3013) to Eligible Patients With Relapsed or Refractory Large B-cell Lymphoma
Brief Title: Expanded Access Program for Epcoritamab
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: GCT3013-101
Record Dates: First submitted 2023-01-23; First posted 2023-02-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Large B-cell Lymphoma; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Primary Mediastinal Large B-cell Lymphoma (PMBCL); High Grade B-cell Lymphoma (HGBCL); Grade 3B Follicular Lymphoma
Keywords: Epcoritamab; GEN3013; Diffuse large B-cell lymphoma; Lymphoma; DuoBody-CD3xCD20; Bispecific antibody; Early access; Double-hit DLBCL; Triple-hit DLBCL; Follicular grade 3b; Transformed DLBCL; High-grade B-cell lymphoma; Primary mediastinal large B-cell lymphoma (PMBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Epcoritamab — Eligible patients will receive epcoritamab (28-day cycle) that will be administered as subcutaneous (SC) injections until disease progression, or one or more of the treatment discontinuation criteria are met.
  Other Names: GEN3013; DuoBody®-CD3xCD20

SUMMARY:
The purpose of this program is to provide investigational epcoritamab, an antibody also known as GEN3013 (DuoBody-CD3xCD20), in an expanded access setting for eligible patients with relapsed and/or refractory (R/R) large B-cell lymphoma (LBCL) who have a high unmet medical need with no other treatment options. It is a requirement that patients do not qualify for an ongoing epcoritamab clinical program or are unable to participate due to logistical reasons.

Access to investigational epcoritamab can be requested by contacting preapprovalaccessprograms@genmab.com.

DETAILED DESCRIPTION:
This is a multicenter program conducted within the United States. The program will consist of screening, treatment (Cycle 1 Day 1 until epcoritamab discontinuation), safety follow-up, post-treatment and/or survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* R/R CD20+ mature B-cell neoplasm
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0, 1, or 2
* ≥ 2 prior lines of antineoplastic therapy, including ≥ 1 anti-CD20 monoclonal antibody (mAb)
* Fluorodeoxyglucose (FDG) positron emission tomography (PET)-avid and measurable disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Patients considering the EAP should have no other available therapeutic option and cannot be eligible for other epcoritamab trials.
* Patients considering the EAP must be located in proximity to a US site given that the EAP is currently available only in the United States.
* Prior to initiating any program-related assessments or procedures, patients (or their legally acceptable representative) must sign an informed consent form (ICF), which indicates the purpose of the program, the procedures required for the program, and confirms the patient's willingness to participate in the program.

Exclusion Criteria:

* Any prior therapy with an investigational bispecific antibody targeting CD3 and CD20
* Prior treatment with CAR-T therapy within 100 days prior to first epcoritamab administration
* Primary central nervous system (CNS) lymphoma or known CNS involvement by lymphoma
* Confirmed history of or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy. Low-dose prednisolone for rheumatoid arthritis or similar conditions is allowed.
* Active hepatitis B or hepatitis C
* Known clinically significant cardiac disease
* Pregnancy or breastfeeding
* Known hypersensitivity to allopurinol or rasburicase

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult